CLINICAL TRIAL: NCT06885047
Title: Implementation and Pilot Testing of a Culturally Centered CBT Protocol for Suicidal Behaviors Among Youth in Mexico City
Brief Title: Culturally Centered CBT Protocol for Suicidal Behaviors Among Youth in Mexico City
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Instituto Nacional de Psiquiatría Ramon de la Fuente Muñiz (Unknown)
Responsible Party: Principal Investigator, Yovanska Duarte-Velez, Associate Professor (Research), Bradley Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2175765-2; R34MH136224 (NIH)
Record Dates: First submitted 2025-02-18; First posted 2025-03-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Suicidal Ideation/Behavior
Keywords: Randomized Controlled Trial; Mexico youth; cultural adaptation; cognitive behavioral therapy
MeSH Terms: conditions — Suicidal Ideation; Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCBT-SB treatment model (Experimental): A culturally centered CBT treatment protocol called Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB)
  Interventions: Behavioral: Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB)
- Treatment as Usual (Active Comparator): Treatment as usual refers to the type of routine treatment that is provided at the hospital setting.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB) — SCBT-SB is a manualized psychosocial treatment protocol developed specifically with and for L/H youth with suicidal ideation and behaviors. Clinician, adolescents, and caregivers' manuals are available in both Spanish and English. SCBT-SB protocol's main conceptual framework and strategies are informed by Cognitive Behavioral Therapy concepts, psychoeducation, and adolescent parenting strategies. The intervention involves individual, caregivers, and family sessions. SCBT-SB, while maintaining the basic principles of CBT, was further developed to include developmental (e.g., identity), and cultural elements of L/H families (e.g., family communication, language). The protocol has two main phases. Phase 1, the Crisis Module, includes nine standard core sessions, and Phase 2, which proposes a flexible number of sessions, focused on the delivery of interchangeable coping skills modules and the acquisition of skills that reduce STB.
  Arms: SCBT-SB treatment model
Behavioral: Treatment as usual — TAU consists of eclectic brief treatments, including some CBT or psychodynamic strategies that are applied with adolescents or in conjunction with the caregiver. In all cases, psychoeducation is provided to adolescents and their caregivers. Occasionally, they may be referred to some family therapy intervention. All treatments are brief therapy, provided by clinical psychologists and are intended to address the cognitive, emotional, and family factors that affect the adequate psychosocial functioning of the adolescent.
  Arms: Treatment as Usual

SUMMARY:
This NIMH R34 award application proposes to conduct an adaptation, implementation, and pilot testing of the culturally centered CBT protocol, the Socio-Cognitive Behavioral Therapy for Suicidal Behaviors (SCBTSB), among suicidal youth in Mexico City, Mexico.

The research plan will (a) culturally adapt and contextualize the SCBT-SB for its implementation in the Mexican public health system, (b) pilot test the protocol through an RCT (SCBT-SB vs TAU; 60 patients and caregivers) and (c) evaluate the implementation process of the SCBT-SB and assess qualitatively possible factors that may promote or hinder its future uptake.

DETAILED DESCRIPTION:
This R34 application proposes to conduct an adaptation, implementation, and pilot testing of the culturally centered CBT protocol, the Socio-Cognitive Behavioral Therapy for Suicidal Behaviors (SCBT-SB), among suicidal youth in Mexico City, Mexico. SCBT-SB is a psychosocial treatment developed with the support of the NIMH specifically for suicidal Hispanic youth. SCBT-SB is available in Spanish, has an established training model, and has yielded promising results in intent to treat analyses in reducing suicide attempts and depressive symptoms in comparison to treatment as usual (TAU). Furthermore, it is the CBT protocol with the most empirical evidence for Latinx youth with suicidal behaviors. SCBT is attuned to the cultural needs of Hispanic suicidal youth in real-world service settings. The "EPIS" implementation framework (Exploration, Preparation, Implementation, and Sustainment) and the Ecological Validity Model (ECV) will guide the SCBT-SB implementation and cultural adaptation into the Mexican culture and mental health system. The study will be conducted in one of the main public hospitals in Mexico City, the Hospital Psiquiatrico Infantil "Dr. Juan N. Navarro". In line with this objective, the following research aims are proposed: Aim 1: Adapt the SCBT-SB for its implementation and pilot testing in the Mexican public health system. An open trial with 10 participants will be completed as part of the adaptation process before the pilot randomized controlled trial (RCT). Aim 2: To conduct a pilot RCT to assess feasibility, acceptability, and treatment effect of SCBT-SB in clinical outcomes versus treatment as usual (TAU). Participants will be 60 youth ages 12-17 admitted to the inpatient units receiving services for suicidal thoughts and behavior (STB). STB and depressive symptoms will be examined at baseline, at hospital discharge (approximately 2 weeks), six-, and 9-months following baseline. Aim 3: To identify organizational/system-level, provider-level, and client factors that may promote or hinder uptake of the new intervention in the public system.

ELIGIBILITY:
Youth Inclusion Criteria:

* ages 12 to 17,
* severe SI, defined as a score of 22 or above on the SIQ-JR or having made a SA or having a suicidal crisis (e.g., threats of attempting suicide) within the last 3 months
* not be engaged in mental health services outside HPIJNN.

Exclusion Criteria:

* having a diagnosis of a psychotic disorder
* having a diagnosis of substance use disorder, rated severe on the DSM-593 (i.e., endorsement of 6 or more symptoms),
* not having sufficient cognitive ability to enter a psychotherapy service (whether reported by the parents or by data in the clinical record)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  Suicidal ideation measured using the Suicide Ideation Questionnaire-Junior (SIQ-JR), a self-report instrument of 15 items that measures severity of suicidal ideation as a continuous variable with established normative, reliability, and validity data for clinical and non-clinical adolescent samples. The minimum score is 0 and the maximum 90. A higher score represents increased severity and frequency of suicidal thoughts.
Depressive symptoms by self-report | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  Level of depressive symptomatology using the Revised Children's Anxiety and Depression Scale-25 (RCADS-25). The RCADS-25 is a 25-item scale that measures levels of anxiety and low mood (e.g. "I feel sad or empty"). The scale has two subscales (Total Anxiety and Total Depression) and an overall score. The Total Depression subscale consists of 10 items. All items assess the frequency of symptoms and are rated on a 4-point Likert scale from "0" (never) to "3" (always). The minimum score for the total depression subscale is 0 and the maximum 30. A higher score means higher level of depressive symptoms. Scoring the RCADS-25 uses converted scores on the total scale and both sub-scales divided into scoring.
Depressive symptoms by self-report | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  Patient Health Questionnaire-9 (PHQ-9) is a depression scale which scores each of the nine major depressive disorder DSM-IV criteria as "0" (not at all) to "3" (nearly every day). The minimum score is 0 and the maximum 27, with higher scores indicating more severe depressive symptoms. It has been validated for use in primary care and it is widely used to monitor the severity of depression symptoms and response to treatment.
Depressive symptoms by clinical interview | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  Depressive symptoms using the Children's Depression Rating Scale-Revised (CDRS-R). The CDRS-R is a 17-item interview assessment of depressive symptoms for school aged children and adolescents, with item rating between 1 (no difficulties) to 5 or 7 (clinically significant difficulties). The minimum raw score is 17 and the maximum 113. A higher score means higher level of depressive symptoms. It has been proposed that a score of ≥40 indicates depressive symptomatology comparable to a diagnosis of depression, whereas a score ≤28 was often used as indicative of remission within trials.

SECONDARY OUTCOMES:
Suicide Attempts | Change from baseline to 6 months, 6 months to 9 months, and baseline to 9 months.
  Actual and interrupted suicide attempts (yes or no) using the Columbia-Suicide Severity Rating Scale (C-SSRS).

CONTACTS AND LOCATIONS:
Overall Officials: Yovanska Duarte-Velez, PhD, Principal Investigator — Brown University Health
Locations (1):
- The Hospital Psiquiatrico Infantil "Dr. Juan N. Navarro", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Basic demographics and outcome measures will be uploaded to the NIMH Data Archive with a data dictionary.
Supporting Information: CSR
Time Frame: Data will be available starting 6 months after main study results publication.
Access Criteria: Researchers with access to the NIMH Data Archive will have access to the uploaded data. Data will also be made available to other researchers by request through a Data Sharing Agreement between institutions and as per NIH data sharing guidelines. The PI will also consult to anyone interested in replicating the intervention and study.

REFERENCES:
- [Background] Duarte-Velez Y, Jimenez-Colon G, Jones RN, Spirito A. Socio-Cognitive Behavioral Therapy for Latinx Adolescent with Suicidal Behaviors: A Pilot Randomized Trial. Child Psychiatry Hum Dev. 2024 Jun;55(3):754-767. doi: 10.1007/s10578-022-01439-z. Epub 2022 Oct 1. PMID 36183051
- [Background] Jimenez-Colon G, Duarte-Velez Y. Raising Children in Different Cultures: Working with Latinx Youth with Suicidal Behaviors and Their Families. R I Med J (2013). 2022 May 2;105(4):31-35. PMID 35476733
- [Background] Duarte-Velez Y, Torres-Davila P, Spirito A, Polanco N, Bernal G. Development of a treatment protocol for Puerto Rican adolescents with suicidal behaviors. Psychotherapy (Chic). 2016 Mar;53(1):45-56. doi: 10.1037/pst0000044. PMID 26928136